CLINICAL TRIAL: NCT03131596
Title: Prevention of Postoperative Adhesion Reformation by Intrauterine Balloon Therapy: a Randomized Controlled Trial
Brief Title: Postoperative Intermittent Intrauterine Balloon Dilatation Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiaoyu Shi, principal investigator, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016FXHEC-KY036
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Intrauterine Adhesion
Keywords: Intrauterine Adhesion; Hysteroscopy; Intrauterine balloon; Reformation; Prevention
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Both surgeons conducting the hysteroscopic surgery and follow-up hysteroscopy were blinded to the patient group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IUB dilatation therapy (Experimental): The patient will have Foley-catheter intrauterine balloon dilatation 2 weeks and 6 weeks after hysteroscopic adhesiolysis. A second-look hysteroscopy will be carried out in the early proliferative phase 4 weeks after the surgery and third-look hysteroscopy will be carried out 8 weeks after the surgery.
  Interventions: Procedure: IUB dilatation therapy
- control group (No Intervention): Patient will not undergo any balloon therapy. A second-look hysteroscopy will be carried out in the early proliferative phase 4 weeks after the surgery and third-look hysteroscopy will be carried out 8 weeks after the surgery.

INTERVENTIONS:
Procedure: IUB dilatation therapy — A Foley catheter (size 14fr) will be prepared by cutting the excess catheter tip protruding beyond the balloon prior to insertion into the uterine cavity. Once the catheter has reached the fundus, 3-4.5mls of saline will be slowly introduced into the balloon under ultrasound guidance, in order to directly visualize the distention of the cavity and division of any intrauterine adhesions, if present.
  Arms: IUB dilatation therapy

SUMMARY:
In this prospective, randomized, controlled study, the investigators wish to determine the efficacy of intrauterine balloon (IUB) dilatation in the prevention of adhesion reformation when compared with the conventional management.

DETAILED DESCRIPTION:
Patients

The patients will be recruited from the Hysteroscopy Center of the Fuxing Hospital, Beijing, China. Before the surgery all patients with suspected Asherman syndrome will undergo preoperative evaluations, including a detailed history of the menstrual pattern, any previous intrauterine surgery, and reproductive history, as well as trans-vaginal ultrasonography. The severity and extent of intrauterine adhesions will be scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version). The inclusion criteria include [1] women aged 18-40 years; [2] moderate to severe intrauterine adhesion (AFS score≥5); [3] first episode of hysteroscopic adhesiolysis in FuXing hospital; [4] written consent obtained; and [5] agreement to have second-look and an optional third-look hysteroscopy. The exclusion criteria include [1] minimal adhesion (AFS score <5) and [2] previous hysteroscopic adhesiolysis in FuXing hospital.

Study Design

After the completion of hysteroscopic adhesiolysis, recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: [1] having a Foley-catheter intrauterine balloon dilatation 2 weeks and 6 weeks after hysteroscopic adhesiolysis; [2] the control group without any additional treatment. A second-look hysteroscopy will be carried out in the early proliferative phase 4 weeks after the surgery and an optional third-look hysteroscopy will be carried out 8 weeks after the surgery.

Power Calculation

On the basis of the results of the two published retrospective cohort studies comparing the balloon and hormone therapy group (control group) in the prevention of adhesion reformation, we estimate that the adhesion reformation rate in the balloon group to be 20% and in the control group to be 45%. Accepting a type 1 error of 0.05, and a type 2 error of 0.10, the number of subjects in each arm of the randomized, controlled trial would be 79. Assuming that the dropout rate to be 20%, the total number of subject to be recruited would be 100 in each arm.

Procedure

Surgical procedure

The surgery will be carried out by one of two experienced hysteroscopic surgeons with the use of a 8.5-mm rigid hysteroscope (Olympus) with 0.9% normal saline infusion under 120-150 mmHg pressure. The procedure will be performed under general anesthesia in a day surgery unit. Ultrasonographic guidance will be routinely used. Once the extent and severity of uterine adhesion has been assessed, the adhesions will be divided with the use of bipolar instrument until normal uterine anatomy is achieved.

Postoperative treatments

All subjects will be treated with oral antibiotics(Cefaclor 0.375 mg twice daily Tianjin Central Pharmaceutical Co Ltd., Tianjin, China.) for 5-7 days. In all cases hormone therapy also began from the day of operation, consisting of estradiol valerate at a dose of 4 mg/d for 21 days, with the addition of dydrogesterone at a dose of 10 mg/d for the last 7 days of the estrogen therapy. After the withdrawal bleed, the hormone therapy was repeated for a further two cycles, i.e. 3 months in total. Second-look hysteroscopy will be carried out in the early proliferative phase, 4 weeks after the initial operation; a third-look hysteroscopy will be carried out 8 weeks after the initial operation. After assessment of the extent and severity of any reformed adhesion, hysteroscopic adhesiolysis will also be carried out at the time of the second-look procedure, if adhesion has recurred. The surgeon who performs the second-look and third-look hysteroscopy will be blinded to the randomization.

IUB dilatation

IUB dilatation therapy will be performed using a Foley catheter(14fr) and according to the methodology published in the literature. This will be prepared by cutting the catheter tip protruding beyond the balloon. Once the catheter has reached the fundus, 3-4.5mls of saline will be slowly infiltrated into the balloon under ultrasound guidance in order to distend the cavity, thereby separating any reformed intrauterine adhesions.

Statistical Analysis

Intention-to-treat analysis was conducted primarily on all outcomes for all randomized subjects. Numerical data with normal distribution were presented as the mean ± standard deviation, whereas data with skewed distribution were presented as the median (interquartile range). The Student t test was used to compare normally distributed data between two groups and paired t test was used to compare normally distributed data within two groups. The Mann-Whitney U test was used to compare data with skewed distribution. Contingency table analysis and the χ2 test were used to compare categorical data. A p value of < 0.05 was considered statistically significant. All statistical analysis was carried out with the use of SPSS 21.0.

Outcome measures

The primary outcome measure was defined as the AFS score at each follow-up, including the adhesion reformation rate, in addition to the menstrual improvement, which was evaluated according to Pictorial Blood Loss Assessment Chart (PBAC) score.

Secondary outcomes included pregnancy rate, miscarriage rate and ectopic rate.

Data processing and analysis

The investigators will ensure the confidentiality of sensitive data by minimizing the number of personnel who handle subject data. In addition, computer data will be encrypted as required to maximize security, while paper documents will be locked in filing cabinets, with only authorized personnel having access to the information.

Ethical considerations

IUB dilatation has been published as a novel technique with no untoward complications identified to date. The procedure will be performed according to the methodology available in the literature and the study has gained approval from the local ethical committee.

Consent

All subjects will be given a detailed explanation of the study and sufficient time to consider their participation. A written consent form will be signed by the patient and retained in the confidential records.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-40 years;
2. moderate to severe intrauterine adhesion (AFS score≥5);
3. no previous history of hysteroscopic adhesiolysis in our hospital;
4. written consent obtained
5. agreement to have second-look and third-look hysteroscopy.

Exclusion Criteria:

1. minimal adhesion (AFS score <5);
2. previous hysteroscopic adhesiolysis in our hospital.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tinchiu Li, Study Chair — Fuxing Hospital,Capital Medical University，China
Locations (1):
- Fu Xing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saravelos SH, Li TC. Ultrasound-guided treatment of intrauterine adhesions in the outpatient setting. Ultrasound Obstet Gynecol. 2017 Aug;50(2):278-280. doi: 10.1002/uog.16218. No abstract available. PMID 27420903
- [Background] March CM. Intrauterine adhesions. Obstet Gynecol Clin North Am. 1995 Sep;22(3):491-505. PMID 8524533
- [Background] ASHERMAN JG. Traumatic intra-uterine adhesions. J Obstet Gynaecol Br Emp. 1950 Dec;57(6):892-6. doi: 10.1111/j.1471-0528.1950.tb06053.x. No abstract available. PMID 14804168
- [Background] ASHERMAN JG. Amenorrhoea traumatica (atretica). J Obstet Gynaecol Br Emp. 1948 Feb;55(1):23-30. doi: 10.1111/j.1471-0528.1948.tb07045.x. No abstract available. PMID 18902559
- [Background] Valle RF, Sciarra JJ. Intrauterine adhesions: hysteroscopic diagnosis, classification, treatment, and reproductive outcome. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 1):1459-70. doi: 10.1016/0002-9378(88)90382-1. PMID 3381869
- [Background] Orhue AA, Aziken ME, Igbefoh JO. A comparison of two adjunctive treatments for intrauterine adhesions following lysis. Int J Gynaecol Obstet. 2003 Jul;82(1):49-56. doi: 10.1016/s0020-7292(03)00030-4. PMID 12834941
- [Background] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Background] Saravelos SH, Jayaprakasan K, Ojha K, Li TC. Assessment of the uterus with three-dimensional ultrasound in women undergoing ART. Hum Reprod Update. 2017 Mar 1;23(2):188-210. doi: 10.1093/humupd/dmw040. PMID 28007752
- [Background] Grimbizis GF, Di Spiezio Sardo A, Saravelos SH, Gordts S, Exacoustos C, Van Schoubroeck D, Bermejo C, Amso NN, Nargund G, Timmermann D, Athanasiadis A, Brucker S, De Angelis C, Gergolet M, Li TC, Tanos V, Tarlatzis B, Farquharson R, Gianaroli L, Campo R. The Thessaloniki ESHRE/ESGE consensus on diagnosis of female genital anomalies. Gynecol Surg. 2016;13:1-16. doi: 10.1007/s10397-015-0909-1. Epub 2015 Nov 4. PMID 26918000
- [Derived] Shi X, Saravelos SH, Zhou Q, Huang X, Xia E, Li TC. Prevention of postoperative adhesion reformation by intermittent intrauterine balloon therapy: a randomised controlled trial. BJOG. 2019 Sep;126(10):1259-1266. doi: 10.1111/1471-0528.15843. Epub 2019 Jul 18. PMID 31207009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 208 patients with moderate to severe (American Fertility Society score ≥ 5) Asherman syndrome who underwent hysteroscopic adhesiolysis were recruited from May 1st,2017 to January 1st,2018.
Pre-assignment Details: 1 patients was excluded follow the criteria strictly and 7 patients declined to participant. In total, 8 patients were excluded before assignment to groups.
Groups:
- IUB Dilatation Therapy: The patient will have a Foley-catheter intrauterine balloon dilatation 2 weeks and 6 weeks after hysteroscopic adhesiolysis. A second-look hysteroscopy was carried out in the early proliferative phase 4 weeks after the surgery and an optional third-look hysteroscopy will carried out 8 weeks after the surgery.
  IUB dilatation therapy: A Foley catheter (size 8-12fr) will be prepared by cutting the excess catheter tip protruding beyond the balloon prior to insertion into the uterine cavity. Once the catheter has reached the fundus, 3-5mls of saline will be slowly introduced into the balloon under ultrasound guidance, in order to directly visualize the distention of the cavity and division of any intrauterine adhesions, if present.
- Control Group: Patient will not undergo any balloon therapy. A second-look hysteroscopy will be carried out in the early proliferative phase 4 weeks after the surgery and an optional third-look hysteroscopy will be carried out 8 weeks after the surgery.
Period: Overall Study
Arm/Group | IUB Dilatation Therapy | Control Group
Started | 100 | 100
Completed | 94 | 97
Not Completed | 6 | 3
Not completed — Protocol Violation | 3 | 3
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: A total of 208 women were assessed for eligibility between May 2017 and December 2017. Of these women, 200 were eligible and randomized. 9 patients did not complete the full protocol, resulting in 94 cases in the balloon group and 97 cases in the control group.
Groups:
- IUB Dilatation Therapy: The patient will have a Foley-catheter intrauterine balloon dilatation 2 weeks and 6 weeks after hysteroscopic adhesiolysis. A second-look hysteroscopy was carried out in the early proliferative phase 4 weeks after the surgery and an optional third-look hysteroscopy will carried out 8 weeks after the surgery.
  IUB dilatation therapy: A Foley catheter (size 14fr) will be prepared by cutting the excess catheter tip protruding beyond the balloon prior to insertion into the uterine cavity. Once the catheter has reached the fundus, 3-4.5mls of saline will be slowly introduced into the balloon under ultrasound guidance, in order to directly visualize the distention of the cavity and division of any intrauterine adhesions, if present.
- Total: Total of all reporting groups
Arm/Group | IUB Dilatation Therapy | Control Group | Total
Number analyzed (Participants) | 94 | 97 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (4.7) | 32.0 (4.4) | 32.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 97 | 191
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 94 | 97 | 191
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
AFS score before operation [Median (Inter-Quartile Range); unit: units on a scale] — The American Fertility Society(AFS) score was used to represent the severity of the intrauterine adhesion. The score range from 0-12 points.
  0 means the uterine cavity is normal without any adhesion. Mild adhesion 1-4, Moderate adhesion 5-8, Severe adhesion 9-12. The higher the score is, the more severe the adhesion is. We measured the score before the patients had hysteroscopic surgery and 8 weeks after the index surgery in order to assess the efficacy of the balloon dilatation therapy in prevention of IUA.
  units on a scale | 10 [6 to 12] | 10 [6 to 12] | 10 [6 to 12]
PBAC score before operation [Mean (Standard Deviation); unit: units on a scale] — The Pictorial Blood Loss Assessment Chart (PBAC) score was used to represent the menstrual flow volume of the patient. The PBAC score is calculated by collecting the patient's pad and observing the degree of staining. The minium value of PBAC score is 0, which means the patient is amenorrhea.The maximum value of PBAC score is 1000. Usually the score is low in patient with intrauterine adhesion(from 0-30 points).
  We measured the score before and 8 weeks after the operation in order to assess if there was any improvement (higher than before) in menstrual flow.
  units on a scale | 19.4 (8.6) | 18.8 (7.8) | 19.1 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adhesion Reformation (American Fertility Society Score of Greater Than 0) 8 Weeks Later After the Index Surgery
Description: The American Fertility Society (AFS) score ranges from 0-12, while represented the severity of the adhesions. Mild 1-4, Moderate 5-8, Severe 9-12. The lower the AFS score is, the better the prognosis the patient is. When the surgery was finished the AFS score should be 0. The reformation of intrauterine adhesions was evaluated by third-look hysteroscopy, if the score was greater than 0, a adhesion reformation was considered.
Time Frame: at 8 weeks post-operation
Population: Intention-to-treat analysis was conducted on all outcomes.
Measure: Count of Participants; unit: Participants
Groups:
- IUB Dilatation Therapy: The patient will have a Foley-catheter intrauterine balloon dilatation 2 weeks and 6 weeks after hysteroscopic adhesiolysis. A second-look hysteroscopy was carried out in the early proliferative phase 4 weeks after the surgery and third-look hysteroscopy will carried out 8 weeks after the surgery.
  IUB dilatation therapy: A Foley catheter (size 14fr) will be prepared by cutting the excess catheter tip protruding beyond the balloon prior to insertion into the uterine cavity. Once the catheter has reached the fundus, 3-4.5mls of saline will be slowly introduced into the balloon under ultrasound guidance, in order to directly visualize the distention of the cavity and division of any intrauterine adhesions, if present.
Arm/Group | IUB Dilatation Therapy | Control Group
Number analyzed (Participants) | 94 | 97
Participants | 21 | 38
Statistical Analysis 1: Comparison: IUB Dilatation Therapy vs Control Group; 200 patients were eligible and randomised in a 1:1 fashion. 9 patients did not complete the full protocol, resulting in 94 cases in the balloon group and 97 cases in the control group included in the final analysis. Intention-to-treat analysis was conducted.The null hypothesis is the percentage of the patients with reformed uterine adhesion in balloon group will less than the percentage of the patients with reformed uterine adhesion in control group. A Chi-squared analysis was used; Test type: Superiority; p = 0.012, Chi-squared — The p-value is not adjusted and a p-value of < 0.05 is considered statistically significant

2. Primary Outcome: The American Fertility Society Score 8 Weeks After Operation
Description: The American Fertility Society(AFS) score of each group was evaluated again at third-look hysteroscopy in order to reflect the efficacy of the treatment. The original AFS score was recorded in baseline characteristics part. The AFS score ranges from 0-12, while represented the severity of the adhesions. Mild 1-4, Moderate 5-8, Severe 9-12. The lower the AFS score is, the better the prognosis the patient is. When the surgery was finished the AFS score score should be 0.
Time Frame: at 8 weeks post-operation
Population: The AFS score of each group was evaluated again after the whole procedure in order to reflect the efficacy of the treatment.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IUB Dilatation Therapy | Control Group
Number analyzed (Participants) | 94 | 97
score on a scale | 0 [0 to 2] | 2 [2 to 4]
Statistical Analysis 1: Comparison: IUB Dilatation Therapy vs Control Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Pictorial Blood Loss Assessment Chart Score 8 Weeks After Operation
Description: The Pictorial Blood Loss Assessment Chart (PBAC) score was used to represent the menstrual flow volume of the patient. The PBAC score was evaluated again at 8 weeks after surgery. A higher PBAC score after hysteroscopic adhesiolysis means a better outcome.The PBAC score of a normal women usually range from 30-100 points.
  The minium value of PBAC score is 0, which means the patient is amenorrhea. The maximum value of PBAC score is 1000.
  We measured the score before and 8 weeks after the operation in order to assess if there was any improvement (higher than before) in menstrual flow.
Time Frame: at 8 weeks post-operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IUB Dilatation Therapy | Control Group
Number analyzed (Participants) | 94 | 97
score on a scale | 51.3 (7.5) | 31.6 (8.1)
Statistical Analysis 1: Comparison: IUB Dilatation Therapy vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Pregnancy Outcome Within 12 Months Follow-up After Third Look Hysteroscopy
Description: number of patients who have pregnancy, miscarriage and ectopic pregnancy within12 months follow-up
Time Frame: within 12 months after third look hysteroscopy(8 weeks post-operation)
Measure: Count of Participants; unit: Participants
Arm/Group | IUB Dilatation Therapy | Control Group
Number analyzed (Participants) | 94 | 97
Participants
  number of pregnancy | 27 | 26
  number of live birth and ongoing pregnancy | 18 | 16
  number of patients have miscarriage | 8 | 9
  number of patients have ectopic pregnancy | 1 | 1
Statistical Analysis 1: Comparison: IUB Dilatation Therapy vs Control Group; Test type: Superiority; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 months
Description: The adverse events in our study were defined as uterine perforation and fluid overload during the operation; severe bleeding after operation or balloon dilatation; infection after operation or balloon dilatation.
Groups:
- IUB Dilatation Therapy: The patient will have Foley-catheter intrauterine balloon dilatation 2 weeks and 6 weeks after hysteroscopic adhesiolysis. A second-look hysteroscopy will be carried out in the early proliferative phase 4 weeks after the surgery and an optional third-look hysteroscopy will be carried out 8 weeks after the surgery.
  IUB dilatation therapy: A Foley catheter (size 14fr) will be prepared by cutting the excess catheter tip protruding beyond the balloon prior to insertion into the uterine cavity. Once the catheter has reached the fundus, 3-4.5mls of saline will be slowly introduced into the balloon under ultrasound guidance, in order to directly visualize the distention of the cavity and division of any intrauterine adhesions, if present.
Arm/Group | IUB Dilatation Therapy | Control Group
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/97
Other Adverse Events (participants affected / at risk) | 0/94 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03131596/Prot_SAP_000.pdf